CLINICAL TRIAL: NCT07295860
Title: A Multicenter Randomized Trial Comparing FANS-Based Flexible Ureteroscopy Versus Suction Mini-Percutaneous Nephrolithotomy for Renal Stones 2-3 cm. The National Innovative Large Egyptian (NILE) Stone Study.
Brief Title: FANS-FURS vs Suction Mini-PCNL for 2-3 cm Renal Stones: A Multicenter Randomized Trial
Acronym: NILE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NILE Stone Study; RP.25.8.1033 (Other: Faculty of medicine, Mansoura University)
Record Dates: First submitted 2025-12-08; First posted 2025-12-22 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-12

CONDITIONS: Stone, Kidney; Stone, Urinary
Keywords: Renal stones; Nephrolithiasis; Urolithiasis; RIRS; FANS; mini-PCNL; Suction technology; Stone-free rate
MeSH Terms: conditions — Kidney Calculi; Urinary Calculi; Nephrolithiasis; Urolithiasis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Participants and surgeons are unblinded due to the nature of surgical interventions. However, postoperative imaging and clinical outcome assessment will be performed by blinded independent assessors."
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- FANS-Based Flexible Ureteroscopy (FURS) (Experimental)
  Interventions: Procedure: FANS-Based Flexible Ureteroscopy (FURS)
- Suction-Assisted Mini-PCNL (Active Comparator)
  Interventions: Procedure: Suction-Assisted Mini-PCNL

INTERVENTIONS:
Procedure: FANS-Based Flexible Ureteroscopy (FURS) — Under general/ spinal anesthesia, patients will be placed in lithotomy position. After guidewire placement, a flexible navigable suction ureteral access sheath (FANS) will be advanced to the renal pelvis. Lithotripsy will be performed using a digital flexible ureteroscope and holmium laser with optimized settings for dusting and fragmentation. Continuous irrigation combined with active suction will enhance visualization and fragment clearance. A double-J stent will be placed post-procedure.
  Arms: FANS-Based Flexible Ureteroscopy (FURS)
Procedure: Suction-Assisted Mini-PCNL — Under general or spinal anesthesia, patients will be placed in the prone position. Percutaneous renal access will be achieved under ultrasound or fluoroscopy guidance using an 18G puncture needle. Tract dilation will be performed up to 16-22 Fr, followed by the insertion of a suction-enabled miniaturized sheath (e.g., ClearPetra or equivalent). A mini-nephroscope will be introduced to visualize and fragment stones using Holmium:YAG fiber laser. Continuous irrigation combined with active negative-pressure suction through the access sheath will facilitate real-time removal of stone dust and fragments while maintaining low intrarenal pressure and clear visualization. A nephrostomy tube or double-J stent will be inserted at the surgeon's discretion.
  Arms: Suction-Assisted Mini-PCNL

SUMMARY:
This multicenter, prospective, randomized clinical trial compares FANS-assisted flexible ureteroscopy (FURS) with suction-assisted mini-percutaneous nephrolithotomy (mini-PCNL) for the treatment of renal stones measuring 2-3 cm. A total of 280 patients will be enrolled across nine tertiary centers and randomized 1:1 to either technique. The primary endpoint is stone-free rate (SFR) at 1 month, assessed by non-contrast CT. Secondary outcomes include operative time, intraoperative complications, postoperative morbidity (Clavien-Dindo), pain scores, hospital stay, reinterventions, and quality of life (EQ-5D-5L). The study aims to provide the first high-quality head-to-head evidence comparing these two modern suction-enhanced technologies, with the goal of defining the optimal minimally invasive approach for medium-sized renal stones.

DETAILED DESCRIPTION:
Aim of the Study

The primary aim of this study is to compare the stone-free rate (SFR) of FANS-assisted flexible ureteroscopy versus suction-assisted mini-percutaneous nephrolithotomy (mini-PCNL) in patients with renal stones measuring 2 to 3 cm. Secondary aims include comparing perioperative outcomes, complication rates, length of hospital stay, and patient-reported quality of life between the two treatment modalities.

Patients and Methods Study Design

This is a prospective, multicenter, randomized, superiority trial. Patients will be recruited from nine high-volume tertiary referral centers. Participants will be randomized in a 1:1ratio to undergo either FANS-based flexible ureteroscopy or suction mini-PCNL using a computer-generated randomization tables, stratified by each center. Allocation concealment will be maintained using sequentially numbered, opaque, sealed envelopes (SNOSE) prepared by an independent person who is not involved in patients' recruitment or treatment. Surgeons and investigators will be blinded to group allocation until the point of intervention.

Ethical Considerations The study protocol will be approved by the Institutional Review Board (IRB) of each participating center. All patients will provide written informed consent before enrollment. The study will be conducted in accordance with the principles of the Declaration of Helsinki.

Patient Evaluation and Recruitment All patients will undergo a standardized preoperative assessment including medical history, physical examination, blood tests (CBC, renal function, coagulation profile), urinalysis, urine culture, and non-contrast CT (NCCT) for stone size, density (HU), and volume assessment. Eligible patients will be screened and enrolled after providing informed consent. Antibiotic prophylaxis will be administered according to European Association of Urology (EAU) guidelines.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥18 years old.
* Single or multiple renal stones measuring 2 -3 cm (diagnosed by NCCT).
* Negative urine culture prior to surgery.
* Suitable for general/spinal anesthesia.
* Signed informed consent.

Exclusion Criteria:

* Active urinary tract infection.
* Anomalous renal anatomy (e.g., horseshoe kidney).
* Severe ureteral strictures preventing retrograde access.
* Coagulopathy or inability to discontinue anticoagulation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 254 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
stone-free rate (SFR) at 1 month postoperatively | 1 month postoperatively
  . SFR will be evaluated using a spiral non-contrast computed tomography (NCCT) scan performed at 1 month after the procedure. Stone-free status will be categorized as no residual or with residual fragments

CONTACTS AND LOCATIONS:
Locations (9):
- Egypt (9):
  - Urology and nephrology center, Al Mansurah, Outside U.S./Canada
  - Alexandria University, Alexandria
  - Assuit University, Asyut
  - Ain Shams University, Cairo
  - Cairo university, Cairo
  - Minya University, Minya
  - Menoufia University, Shibīn al Kawm
  - Tanta University, Tanta
  - Zagazig university, Zagazig